CLINICAL TRIAL: NCT02179580
Title: A Randomized Double Blind Placebo Control Study of Xiang-Sha-Liu-Jun-Zi-Tang (XSLJZT)in Patients With Irritable Bowel Syndrome
Brief Title: A Study of Xiang-Sha-Liu-Jun-Zi-Tang in Patients With Irritable Bowel Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH103-REC2-016
Record Dates: First submitted 2014-05-27; First posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: Traditional Chinese Medicine; Clinical trial; Good Clinical Practice
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xiang-Sha-Liu-Jun-Zi-Tang (Experimental): Xiang-Sha-Liu-Jun-Zi-Tang at a rate of 3.0 g three times per day for 28 days
  Interventions: Drug: Xiang-Sha-Liu-Jun-Zi-Tang; Drug: Placebo
- Placebo (Placebo Comparator): Placebo at a rate of 3.0 g three times per day for 28 days
  Interventions: Drug: Xiang-Sha-Liu-Jun-Zi-Tang; Drug: Placebo

INTERVENTIONS:
Drug: Xiang-Sha-Liu-Jun-Zi-Tang — Xiang-Sha-Liu-Jun-Zi-Tang at a rate of 3.0 g three times per day for 28 days. We use the Chinese herb for the treat of IBS patient
Drug: Placebo — Xiang-Sha-Liu-Jun-Zi-Tang at a rate of 3.0 g three times per day for 28 days. Placebo drug is 1/10 dose of experiment drug .

SUMMARY:
Ministry of Health and Welfare Department of Chinese Medicine and pharmacy specially subsidizes domestic teaching hospitals to install clinical study centers for Chinese pharmacies, in order to establish the clinical study environment for Chinese pharmacies meeting the international regulations, to assist promoting and performing clinical studies in Chinese pharmacies, and then to improve the nation's health and benefits. This will render Chinese pharmacies competitive in the international market by employing scientific tests and verifications. The new project applications are respectively as follows: A randomized double blind placebo control study of Xiang-Sha-Liu-Jun-Zi-Tang (XSLJZT) in patients with irritable bowel syndrome The main clinical manifestations of irritable bowel syndrome (IBS) are chronic, recurrent abdominal pain or abdominal dyscomfortable associated with the changes of defecation habit, such as constipation and/or diarrhea. Clinical treatment of IBS includes behavioral, and drug treatment, such as anti-diarrheal agent, 5-HT3 receptor antagonist and 5-HT4 receptor agonist, but these treatments relieve partial symptoms only. Xiang-Sha-Liu-Jun-Zi-Tang (XSLJZT) origins from Yizongjinjion, and that uses XSLJZT to treat the patients who has qi deficiency, phlegm-retained fluid, nausea and vomiting, gastrointestinal dysharmony and producing many symptoms. These symptoms of mentioned-above are similar to IBS. Therefore, the purpose of the present study was to investigate the therapeutic effect of XSLJZT on IBS, the investigators designed a randomized double blind placebo control study to assess the effect of XSLJZT on IBS.

DETAILED DESCRIPTION:
Ministry of Health and Welfare Department of Chinese Medicine and pharmacy specially subsidizes domestic teaching hospitals to install clinical study centers for Chinese pharmacies, in order to establish the clinical study environment for Chinese pharmacies meeting the international regulations, to assist promoting and performing clinical studies in Chinese pharmacies, and then to improve the nation's health and benefits. This will render Chinese pharmacies competitive in the international market by employing scientific tests and verifications. The new project applications are respectively as follows: A randomized double blind placebo control study of Xiang-Sha-Liu-Jun-Zi-Tang (XSLJZT) in patients with irritable bowel syndrome The main clinical manifestations of irritable bowel syndrome (IBS) are chronic, recurrent abdominal pain or abdominal dyscomfortable associated with the changes of defecation habit, such as constipation and/or diarrhea. Clinical treatment of IBS includes behavioral, and drug treatment, such as anti-diarrheal agent, 5-HT3 receptor antagonist and 5-HT4 receptor agonist, but these treatments relieve partial symptoms only. Xiang-Sha-Liu-Jun-Zi-Tang (XSLJZT) origins from Yizongjinjion, and that uses XSLJZT to treat the patients who has qi deficiency, phlegm-retained fluid, nausea and vomiting, gastrointestinal dysharmony and producing many symptoms. These symptoms of mentioned-above are similar to IBS. Therefore, the purpose of the present study was to investigate the therapeutic effect of XSLJZT on IBS, we designed a randomized double blind placebo control study to assess the effect of XSLJZT on IBS.

In addition to the performance of the clinical study projects for Chinese pharmacies, our center will still maintain cooperation with domestic or foreign biotechnology industries, the industries of Chinese herbal medicine and academic research institutes, such as the material research institute in Industrial Technology Research Institute, Feng Chia University, and Yuanpei University, make efforts in expanding the study in the development of novel Chinese medicinal drugs and novel medical techniques, and cooperate with famous international Contract Research Organizations (CRO). We want to build a clinical study service platform, in which the internal part is to integrate various R&D units on campuses and hospitals, such as the teams in the department of medical care, department of medical technology, all laboratories, the incubation center, the biostatistics center, the administrative department and improve the internal procedures for performing clinical studies. The external part is to make efforts to win over domestic and foreign clinical study cases to be performed in our center. The performing methods are illustrated as follows:

1. Setting up the environment and related equipment that enable the performance of clinical studies in Chinese pharmacies and establishing the operation manuals and standard operation procedures for performing the R&D stage for drugs of Chinese pharmacies.
2. Employing professionals required in the clinical study in Chinese pharmacies and encouraging doctors, pharmacists and nurses to attend advanced study and receive training while enhancing the incubation for the required professionals of clinical studies, such that the experience can be passed to others.
3. Practically performing one or more proposals of developing new drugs of Chinese pharmacies or the clinical study proposal of reassessing therapeutic efficacies of drugs in the drug permission certificates issued by the Committee on Chinese Medicine and Pharmacy on record.
4. Promoting and building an intact and strong audit system in accordance with Good Clinical Practice (GCP), elevating the clinical study level in our country, and putting the regulations of GLP into practice.
5. Promoting the cooperation with industries, academics, and governments and international cooperation.

ELIGIBILITY:
Inclusion Criteria:

1. Age : from 20 y/o to 65 y/o.
2. Gender : male or female.

Exclusion Criteria:

1. Pregnant or lactating.
2. Elevated serum ALT / AST level (3 x upper limit of normal (ULN)),or greater than normal serum Creatinine.
3. The clients with psychological cannot cooperate with each other. ( ex. depression, schizophrenia )
4. Abdominal surgery.
5. Major medical diseases. ( ex. heart failure, myocardial infarction, chronic obstructive pulmonary disease, kidney failure, cancer, stroke )
6. The patient refused to sign informed consent form.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal System Rating Scale-IBS Questionnaire | Change from baseline Gastrointestinal System Rating Scale-IBS score at week 4 (28 ± 5 days) and week 12 (84 ± 7 days)

SECONDARY OUTCOMES:
IBS-QOL Questionnaire | Change from baseline IBS-QOL score at week 4 (28 ± 5 days) and week 12 (84 ± 7 days)

OTHER OUTCOMES:
WHO Quality Questionnaire | Change from baseline WHO Quality of Life-BREF score at week 4 (28 ± 5 days) and week 12 (84 ± 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Hsuehchou Lai, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan